CLINICAL TRIAL: NCT05956873
Title: Multi-center Study on the Endovascular Aortic Repair of Free and Contained Ruptured Thoraco-Abdominal Aortic Aneurysm
Brief Title: Endovascular Aortic Repair of Free and Contained Ruptured Thoraco-Abdominal Aortic Aneurysm
Acronym: REVAR-TAAA
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Enrico Gallitto, MD, PhD, FEBVS, University of Bologna
Other Study IDs: REVAR-TAAA
Record Dates: First submitted 2023-07-01; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Thoracoabdominal Aortic Aneurysm; Ruptured Thoracic Aneurysm; Ruptured Aortic Aneurysm; Thoracoabdominal Aortic Aneurysm, Ruptured
Keywords: Ruptured Thoracoabdominal aortic aneurysm; fenestrated endovascular repair; branched endovascular repair; contained rupture aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal; Aortic Rupture; Rupture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- RTAAA patients treated with REVAR: Included population were consecutive patients presented with evidence of active bleeding (frank ruptures), or without active bleeding but with periaortic structures infiltration/hematoma (contained rupture); undergoing urgent/emergent endovascular RTAAA (Crawford's extend I-IV + suprarenal AAA) repair within the first 24 hours, requiring a proximal landing zone above the celiac trunk with off-the-shelf, F/B-EVAR, PMEG and PG.
  Interventions: Device: REVAR

INTERVENTIONS:
Device: REVAR — Endovascular repair of ruptured TAAAs with available technique and devices: endovascular treatments were performed in urgent or emergent setting, compulsory within the first 24 hours, using an off-the-shelf stent grafts, or an available custom-made fenestrated/branched device or a physician-modified endografts with fenestrations/branches or parallel endografting for renal and visceral arteries

SUMMARY:
Ruptured thoracoabdominal aortic aneurysm (TAAA) represents an emergency medical challenge that needs to be treated promptly. Over the past years different endovascular techniques have emerged such as fenestrated or branched endovascular aortic repair (FB-EVAR). However, FB-EVAR is a technique that uses a custom-made device which needs to be manufactured and this process take months, therefore, it could not be used in urgent settings. Off-the-shelf graft stents are pre-made graft stents, which can be used in urgent cases.

A retrospective, multicenter cohort study was planned to include patients who underwent endovascular procedures between January 2015 and January 2022 (85 months) to evaluate the technical and survival outcomes of the use of off-the-shelf stent graft, physician-modified endograft and parallel graft technique in endovascular aortic repair of free and contained ruptured TAAA.

Data will be collected anonymously and retrospectively, including patient demographics, risk factors, diagnosis and anatomical details, procedure details and post-operative outcomes.

DETAILED DESCRIPTION:
The presentation of a thoracoabdominal aortic aneurysm (TAAA) represents a major clinical challenge leading to a high risk of mortality Traditional open surgical repair has a perioperative mortality risk of 53% and therefore a less invasive option is mandatory. Endovascular abdominal aortic repair (EVAR) has been proposed as the main alternative treatment to reduce mortality compared to open surgical repair, with an advantage of decreasing the risk for renal and pulmonary complications. Over the last two decades, fenestrated and branched EVAR (FB-EVAR) have been implemented as an emerging endovascular techniques for patients with complex abdominal aortic aneurysms to preserve visceral and renal arteries.

FEVAR is a technique using a custom-made device, which requires a production and delivery time of about 90 days and therefore could not be used in urgent settings. However, in urgent cases off-the-shelf stent grafts have been used as alternative options, with a 30-day mortality of 14%. In these settings, and both early and follow-up survival outcomes are strongly affected by hemodynamic patient presentation that represents a main prognostic factor Nonetheless, in urgent cases in whom off-shelf stent grafts cannot be implanted due to complex anatomical configuration, physician-modified endografts (PMEG) have been proposed with an early survival rate ranging from 8% to 14%.

Parallel grafts can be used as a third option, with a comparable overall mortality but with a 24% risk of developing type Ia endoleak, without a complete exclusion of the aneurysmal sac.

Many papers consider free ruptures, contained symptomatic ruptures as well as large aneurysm (diameter >80 with a high risk of ruptures) as an urgent TAAA, but since the hemodynamic status and the symptoms presentation may be strongly different, they should be addressed separately and large-number paper with the focus specifically or ruptured TAAA are still lacking Currently, off-the-shelf stent grafts, PMEG and parallel grafts have been used in many centers across the world for the treatment of ruptured and symptomatic contained ruptured TAAA. Therefore, performing a multicenter study analyzing the data collected may lead to a better understanding of the clinical features as well as the used techniques, outcomes and applicability.

AIMS OF THE STUDY A retrospective multicenter, cross-sectional cohort study to evaluate the technical and survival outcomes of the use of off-the-shelf graft stent, physician-modified-endografts and parallel grafts in endovascular aortic repair of free ruptured and contained ruptured TAAA.

Results and postoperative events will be reported following the current reporting standards for endovascular aortic repair prepared and revised by the Ad Hoc Committee for Standardized Reporting Practices in Vascular Surgery of The Society for Vascular Surgery/American Association for Vascular Surgery.

ELIGIBILITY:
Inclusion Criteria:

Age: Adults Gender: Male and Female Diagnosis of TAAA (Crawford I-V), penetrating aortic ulcers, or failure of previous EVAR, which require proximal landing zone above the celiac trunk. Different etiologies will be accepted with similar anatomical extend (degenerative, post-dissection, inflammatory, etc.) Free and contained ruptured TAAA confirmed by pre-operative computed tomography angiography (CTA).

Patient presenting with and without hemodynamic instability. A free-rupture is considered an aortic rupture with evidence of bleeding outside the aortic wall.

A contained rupture is considered if the integrity of the aortic wall is lots, without clear evidence of bleeding, but with periaortic structures imbibition and periaortic hematoma.

Hemodynamic instability is defined as the presence of cardiopulmonary arrest or the inability to achieve or to maintain a systolic blood pressure > 90 mmHg despite appropriate fluid resuscitation.

Exclusion Criteria:

Patients treated with open or hybrid repair. Patients with TAAA without any sign of aortic wall rupture or without pre-operative CTA.

Patient with contained rupture presenting with no symptoms and discovered accidentally Patient that were transferred to normal wards in the period from diagnosis to procedure or can be treated in elective setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included were all treated for rupture TAAAs in urgent setting using an off-the-shelf stent grafts, or a custom made available fenestrated and branched device, or a physician-modified endografts with fenestrations/branches or in-situ laser fenestration or parallel endografting for renal and visceral arteries.
  o An urgent procedure that is carried out immediately after patient admission or within the first 24-hours.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of Technical Success | Within first post-operative day
  successful endovascular access and deployment of all devices at the intended aortic location, successful catheterization and stenting of all planned target vessels, absence of type I /III endoleaks at the final angiography. The presence of hemodynamic instability at the end of procedure with evidence of bleeding and intra-operative mortality without possibility of completing the procedure, were considered technical failures.
Rate of early mortality | Within 30-days from the procedure.
  We considered as a cumulative endpoint composed by perioperative mortality (within the first 48hours), 30-day Mortality, if the patient died in the first 30-day period after intervention and In-hospital mortality, if the patient died in-hospital with hospitalization time longer than 30-days.
Rate of overall survival | Within 60-months from the procedure
  Overall survival regardless the aortic relationship of the reported cause of death.

SECONDARY OUTCOMES:
Rate of Major Adverse events (MAEs) and rate early re interventions | Within 30-days from the procedure.
  cardiac complications (including myocardial infarction, congestive heart failure, and myocardial ischemia requiring intervention); respiratory complications (including required prolonged >24 hours mechanical ventilation or respiratory insufficiency/pneumonia requiring reintubation and/or ventilatory assistance); acute kidney injury, defined as renal function decline resulting in >30% reduction in baseline eGFR or new-onset dialysis; major stroke, defined as the presence of invalidting neurological sequelae; spinal cord ischemia (SCI) defined as the presence of paraplegia or paraparesis, being temporary if had a complete resolution and expected return to baseline, and permanent if the injury had partial or no improvement compared with baseline examination; bowel ischemia requiring surgical resection or not resolving with medical therapy;
rate of freedom from reintervention | Within 60-months from the procedure
  Overall freedom from need for re interventions related in some extend to the REVAR procedure or RTAAAs condition

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: Undecided
This study is a multicenter, observational, cross-sectional cohort study to evaluate the outcomes of endovascular aortic repair of symptomatic contained and free ruptured TAAAs using off-the-shelf stent grafts and physician-modified stent grafts.
  The study will be a multicenter retrospective cohort including international centers.
  As soon as we receive positive answers from the invited centers, we will proceed to update the protocol, accordingly.

REFERENCES:
- [Background] Locham SS, Grimm JC, Arhuidese IJ, Nejim B, Obeid T, Black JH 3rd, Malas MB. Perioperative Outcomes of Open versus Endovascular Repair for Ruptured Thoracoabdominal Aneurysms. Ann Vasc Surg. 2017 Oct;44:128-135. doi: 10.1016/j.avsg.2017.02.015. Epub 2017 May 10. PMID 28501656
- [Background] Oderich GS, Forbes TL, Chaer R, Davies MG, Lindsay TF, Mastracci T, Singh MJ, Timaran C, Woo EY; Writing Committee Group. Reporting standards for endovascular aortic repair of aneurysms involving the renal-mesenteric arteries. J Vasc Surg. 2021 Jan;73(1S):4S-52S. doi: 10.1016/j.jvs.2020.06.011. Epub 2020 Jun 29. PMID 32615285
- [Background] Spath P, Tsilimparis N, Furlan F, Hamwi T, Prendes CF, Stana J. Additional Aortic Coverage With an Off The Shelf, Multibranched Endograft Compared With Custom Made Devices For Endovascular Repair of Pararenal Abdominal Aortic Aneurysms. Eur J Vasc Endovasc Surg. 2023 May;65(5):710-718. doi: 10.1016/j.ejvs.2023.01.030. Epub 2023 Jan 24. PMID 36707021
- [Background] Gallitto E, Faggioli G, Spath P, Pini R, Mascoli C, Logiacco A, Gargiulo M. Urgent endovascular repair of thoracoabdominal aneurysms using an off-the-shelf multibranched endograft. Eur J Cardiothorac Surg. 2022 May 2;61(5):1087-1096. doi: 10.1093/ejcts/ezab553. PMID 34964451
- [Background] Gallitto E, Faggioli G, Spath P, Pini R, Mascoli C, Ancetti S, Stella A, Abualhin M, Gargiulo M. The risk of aneurysm rupture and target visceral vessel occlusion during the lead period of custom-made fenestrated/branched endograft. J Vasc Surg. 2020 Jul;72(1):16-24. doi: 10.1016/j.jvs.2019.08.273. Epub 2020 Feb 13. PMID 32063442
- [Background] Tsilimparis N, Gouveia E Melo R, Schanzer A, Sobocinski J, Austermann M, Chiesa R, Resch T, Gargiulo M, Timaran C, Maurel B, Adam D, Dias N, Oderich GS, Kolbel T, Gomez Palones F, Simonte G, Giudice R, Mesnard T, Loschi D, Leone N, Gallito E, Spath P, Porras Colon J, Elboushi A, Wachtmeister M, Sonesson B, Tenorio E, Panuccio G, Isernia G, Bertoglio L. Transatlantic multicenter study on the use of a modified preloaded delivery system for fenestrated endovascular aortic repair. J Vasc Surg. 2023 Oct;78(4):863-873.e3. doi: 10.1016/j.jvs.2023.05.043. Epub 2023 Jun 16. PMID 37330705
- [Background] Tsilimparis N, Bosiers M, Resch T, Torsello G, Austermann M, Rohlffs F, Coates B, Yeh C, Kolbel T. Two-year target vessel-related outcomes following use of off-the-shelf branched endografts for the treatment of thoracoabdominal aortic aneurysms. J Vasc Surg. 2023 Aug;78(2):289-298. doi: 10.1016/j.jvs.2023.03.498. Epub 2023 Apr 11. PMID 37044318
- [Derived] Spath P, Tsilimparis N, Gallitto E, Becker D, Vacirca A, Berekoven B, Panuccio G, Karelis A, Kahlberg A, Melissano G, Dias N, Kolbel T, Austermann M, Faggioli G, Oderich G, Gargiulo M; International Collaborators writing committee on TAAA ruptures' study group. Endovascular Repair of 100 Urgent and Emergent Free or Contained Thoracoabdominal Aortic Aneurysms Ruptures. An International Multicenter Trans-Atlantic Experience. Ann Surg. 2025 Mar 1;281(3):522-531. doi: 10.1097/SLA.0000000000006231. Epub 2024 Feb 7. PMID 38323417